CLINICAL TRIAL: NCT01464866
Title: Effect of Nutritional Supplementation on Pediatric Burn Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BK56
Record Dates: First submitted 2011-11-01; First posted 2011-11-04 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2011-11

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Dietary Supplements; Food Service, Hospital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hospital Feed (Active Comparator): Standard hospital food
  Interventions: Other: Hospital food
- Hospital Feed plus nutritional supplement (Experimental): Standard hospital food plus nutritional supplement
  Interventions: Other: Nutritional Supplement

INTERVENTIONS:
Other: Nutritional Supplement — Liquid, pediatric nutritional supplement. 1-2 bottles/day for up to 28 days.
  Arms: Hospital Feed plus nutritional supplement
Other: Hospital food — Typical hospital food given daily at meals
  Arms: Hospital Feed

SUMMARY:
This study will determine the effect of nutrition supplementation on blood protein levels in pediatric burn patients.

ELIGIBILITY:
Inclusion Criteria:

1. 1-10 years of age
2. Hospital admission within 24 hours post-burn
3. At least 15% TBSA burned to at least 2nd degree and no more than 5% TBSA 4th degree or higher
4. Capable of exclusive oral feeding within 3 days of hospitalization
5. Expected to be hospitalized at least 14 days

Exclusion Criteria:

1. History diabetes or stress-induced hyperglycemia
2. Artificial ventilation
3. Requires parenteral or enteral feeding
4. IV albumin
5. Drug that affects metabolism
6. Receiving Dialysis
7. Acutely impacted or constipated
8. Consumes non-study nutritional supplement
9. Allergy or intolerance to any study product ingredient
10. Participating in non-Abbott approved concomitant trial

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2010-02; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
prealbumin | Change between Baseline and Day 14

SECONDARY OUTCOMES:
Preablumin | Change between Baseline and Day 7
C Reactive Protein (CRP) | Between baseline and Day 7
C Reactive Protein | Between baseline and Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Williams, MPH, Study Chair — Abbott Nutrition
Locations (9):
- Russia (9):
  - First Republic Clinical Hospital of Ministry of Healthcare of Udmurtia Republic, Izhevsk
  - Children's Republican Clinical Hospital of Ministry of Healthcare of Tatarstan Republic, Kazan'
  - City Clinical Hospital #2, Kemerovo
  - Children's City Hospital #9, Moscow
  - Nizhny Novgorod Research Institute of Traumatology & Orthopedics of Federal Agency of High Technology Medical Care, Nizhny Novgorod
  - City Hospital #20, Rostov-on-Don
  - Children's City Hospital #1, Saint Petersburg
  - City Clinical Hospital #7, Saratov
  - Children City Clinical Hospital #9, Yekaterinburg